CLINICAL TRIAL: NCT06729281
Title: The Effect of Kinesio Taping on Posture in Healthy Young Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elem Yorulmaz (Other)
Responsible Party: Sponsor-Investigator, Elem Yorulmaz, Doctor academic member, Haydarpasa Numune Training and Research Hospital
Organization: Haydarpasa Numune Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-62977267-903.99-23331179
Record Dates: First submitted 2024-11-21; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Healthy Young Adults Who Are Health Care Workers at Haydarpaşa Numune Training and Research Hospital
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise (No Intervention): Regular exercise is also among the factors affecting the formation of posture. A regular and systematic exercise program can change the curvatures of the spine in the sagittal plane.
- exercise and kinesio taping (Other): Regular exercise is also among the factors affecting the formation of posture. A regular and systematic exercise program can change the curvatures of the spine in the sagittal plane. + Kinesiotaping
  Interventions: Device: kinesio tape

INTERVENTIONS:
Device: kinesio tape — The application of kinesio tape is a relatively new method, first developed in 1973 by Kenzo Kase in Japan, also known as elastic bandage, which has become popular in the last 10 years following announcements at major events such as the Olympic Games.
  Arms: exercise and kinesio taping

SUMMARY:
Healthy young adults who are health care workers at Haydarpasa Numune Training and Research Hospital will be included in the study considering the inclusion and exclusion criteria. Demographic data such as age, gender, height, weight will be recorded. Thoracic kyphosis and lumbar lordosis angles of the participants will be recorded with Goniometer pro application at the beginning. Spinal muscle thickness including the back extensor muscle group will be measured from the thoracic and lumbar regions with ultrasound by a specialist with clinical experience for ultrasound. Measurement will be made at T8 level for thoracic region and L3 level for lumbar region. They will be evaluated with the Nottingham health profile.

A total of 78 people will be included in the study and will be randomly divided into two groups as intervention + exercise and exercise only group. Randomization will be done by closed envelope method. Kinesiobanting will be applied to the intervention group for 4 weeks, with the posture correction technique on Mondays, and the kinesiobant application will be applied once a week for 4 sessions in total, to be removed on Friday. Both groups will be given a 40-minute posture exercise program based on clinical experience, to be performed every other day, i.e. 4 times a week for 12 weeks. Patients will be given an exercise follow-up chart and will be called once a week and followed up for 12 weeks. In the intervention group, thoracic kyphosis and lumbar lordosis angle measurements with Goniometer pro application will be examined at 30.minute at baseline, Week 4 and Week 12, while in the exercise only group they will be examined at baseline, Week 4 and Week 12. Ultrasound measurement of spinal muscle thickness will be performed at baseline and at Week 12 in both groups. Nottingham Health Profile will be performed at baseline, Week 4 and Week 12 in both groups. Differences within and between groups will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Health workers
* Over 18 and under 40
* Visual analog scale (VAS) < 4 for muscle pain
* Inactive (category 1) and minimally active (category 2) according to the international physical activity survey
* Healthcare workers without cognitive deficits who can take verbal instructions

Exclusion Criteria:

* Diagnosed disc herniation with or without spinal deformity
* Bone abnormality and peripheral symptoms
* Infectious or inflammatory arthropathies
* History of joint replacement surgery,
* History of spinal surgery
* Need for assistive devices for ambulation
* irregular hypertension
* Uncontrolled diabetes mellitus
* Presence of neurological disease
* History of malignancy
* Uncontrolled cardiopulmonary disease
* Pregnancy
* Morbid obesity (Body mass index > 35)
* Having fibromyalgia syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Thoracic kyphosis and lumbar lordosis measurements with Goniometer Pro Application | 1. month and 3. month
  Thoracic kyphosis and lumbar lordosis angle measurements with Goniometer pro application will be examined at 30 minutes at baseline, Week 4 and Week 12, whereas only in the exercise group will be examined at baseline, Week 4 and Week 12.
Spinal muscle thickness measurements with Ultrasound | 1. month and 3. month
  Ultrasound measurement of spinal muscle thickness will be performed with Mindray brand ultrasound in both groups at baseline and at week 12, with measurements indicated in millimetres.

SECONDARY OUTCOMES:
Nottingham Health Profile | 1.month and 3. month
  Nottingham Health Profile will be performed at baseline, Week 4 and Week 12 in both groups. Differences within and between groups will be analyzed statistically

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpaşa Numune Training and Research Hospital Physical Medicine and Rehabilitation Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pai S A, Zhang H, Shewchuk JR, Al Omran B, Street J, Wilson D, Doroudi M, Brown SHM, Oxland TR. Quantitative identification and segmentation repeatability of thoracic spinal muscle morphology. JOR Spine. 2020 Jul 1;3(3):e1103. doi: 10.1002/jsp2.1103. eCollection 2020 Sep. PMID 33015576